CLINICAL TRIAL: NCT02932982
Title: Diagnostic Reasoning and Sense of Alarm at Dyspnoea and / or Chest Pain
Acronym: RaisDiag
Status: Terminated | Type: Observational
Why Stopped: No more patients to include
Sponsor: University Hospital, Brest (Other)
Collaborators: University of Anvers (Unknown); Ecole doctorale de Bretagne en biologie de santé (Unknown)
Responsible Party: Sponsor
Other Study IDs: 29BRC16.0143
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Chest Pain; Dyspnea
Keywords: primary care; chest pain; dyspnea
MeSH Terms: conditions — Chest Pain; Dyspnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Dyspnea and chest pain represent 1.5% of general practice consultations. They may be a sign of many diseases, potentially serious. The concept of Gut Feelings brings a sense of alarm and reinsurance. The sense of alarm reflects a sense of mistrust about the patient's clinical situation, in the absence of objective argument. The sense of reinsurance reflects a sense of confidence about the patient's situation, in the absence of objective argument. Gut Feelings plays a key role in the diagnostic reasoning in general practice. A questionnaire measuring the Gut Feelings was validated in French after a linguistic validation procedure.

DETAILED DESCRIPTION:
Dyspnea and chest pain represent 1.5% of general practice consultations. They may be a sign of many diseases, potentially serious. The concept of Gut Feelings brings a sense of alarm and reinsurance. The sense of alarm reflects a sense of mistrust about the patient's clinical situation, in the absence of objective argument. The sense of reinsurance reflects a sense of confidence about the patient's situation, in the absence of objective argument. Gut Feelings plays a key role in the diagnostic reasoning in general practice. A questionnaire measuring the Gut Feelings was validated in French after a linguistic validation procedure.

The objective of the research is to calculate the precision of the sense of alarm the general practitioner facing a consultant for chest pain or dyspnea and patient

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years
* Patients consulting on primary care for chest pain or dyspnea

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 80 years and consulting on primary care for chest pain or dyspnea
Sampling Method: Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
calculate the accuracy of the sense of alarm the general practitioner face a patient consultant for chest pain or dyspnea. | 4 weeks
  Questionary

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - LE GOFF Delphine, La Forêt Landerneau, France
  - ABALAIN-VOREUX Aurélie, Brest
  - SIMON Benjamin, Brest
  - AUFFRET Jean François, Camaret-sur-Mer
  - POINOT Anne, Guerlesquin
  - BEURTON-COURAUD Lucas, Pleyben
  - LE DUFF Nicolas, Ploudalmézeau
  - BODIN Bénédicte, Plounéour-Trez
  - CAM Françoise, Plouzané
  - LOSQUIN André, Pont-l'Abbé
  - MAHE Gwénaëlle, Saint-Nicolas-du-Pélem

REFERENCES:
- [Derived] Barais M, Fossard E, Dany A, Montier T, Stolper E, Van Royen P. Accuracy of the general practitioner's sense of alarm when confronted with dyspnoea and/or chest pain: a prospective observational study. BMJ Open. 2020 Feb 18;10(2):e034348. doi: 10.1136/bmjopen-2019-034348. PMID 32075841